CLINICAL TRIAL: NCT02478008
Title: A Clinical Study of the CardiAQ™ Transcatheter Mitral Valve Implantation (TMVI) System (Transapical Delivery System)
Brief Title: A Clinical Study of the CardiAQ™ TMVI System (Transapical DS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Edwards acquired CardiAQ and opted to terminate this study. 2 patients were enrolled and follow-up is complete. No further enrollment or follow-up will occur.
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-3102-01
Record Dates: First submitted 2015-06-17; First posted 2015-06-23 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2015-09

CONDITIONS: Mitral Insufficiency; Heart Valve Disease; Cardiovascular Disease; Heart Disease
Keywords: Transcatheter Mitral Valve Replacement; Mitral Regurgitation; Mitral Insufficiency; Transapical
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Valve Diseases; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CardiAQ TMVI System (Transapical DS) (Experimental)
  Interventions: Device: CardiAQ TMVI System (Transapical DS)

INTERVENTIONS:
Device: CardiAQ TMVI System (Transapical DS)

SUMMARY:
The purpose of the study is to evaluate the initial short and long-term safety and performance of the CardiAQ™ Transcatheter Mitral Valve Implantation System using the Transapical Delivery System.

The study will enroll patients with moderate to severe mitral valve regurgitation who are considered high or extreme risk for mortality and morbidity from conventional open heart surgery.

ELIGIBILITY:
Key Inclusion Criteria:

* NYHA Classification ≥ III
* Left Ventricular Ejection Fraction ≥ 30%
* Mitral regurgitation ≥ Grade 3+
* Subject meets anatomical eligibility criteria for the investigational device

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Composite Major Adverse Event Rate | 30-Day
Composite Major Adverse Event Rate | 12-Month

CONTACTS AND LOCATIONS:
Overall Officials: Lars Søndergaard, MD, DMSc, Principal Investigator — Rigshospitalet University Hospital (Copenhagen, Denmark)
Locations (9):
- Rigshospitalet University Hospital, Copenhagen, Denmark
- France (3):
  - Centre hospitalier régional universitaire de Lille, Lille
  - Hôpital Européen Georges-Pompidou, Paris
  - Centre Hospitalier Universiatier de Toulouse, Toulouse
- Netherlands (3):
  - Medisch Centrum Leeuwarden, Leeuwarden
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus University Medical Center, Rotterdam
- United Kingdom (2):
  - Leeds General Infirmary, Leeds
  - New Cross Hospital Heart Center, Wolverhampton